CLINICAL TRIAL: NCT00640146
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo Controlled Phase 2 Study of Once-Daily Subcutaneous Methylnaltrexone (MNTX) in the Treatment of Opioid-Induced Constipation During Rehabilitation After Orthopedic Procedures
Brief Title: Study of Subcutaneous Methylnaltrexone (MNTX) in the Treatment of Opioid-Induced Constipation During Rehabilitation After Orthopedic Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNTX2101
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Opioid-induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MNTX (Experimental): Participants will receive methylnaltrexone (MNTX) 12 milligrams (mg) subcutaneously (SC) once daily for up to 4 or 7 days, depending upon the protocol version under which each participant is enrolled.
  Interventions: Drug: Methylnaltrexone bromide
- Placebo (Placebo Comparator): Participants will receive placebo matching to MNTX SC once daily for up to 4 or 7 days, depending upon the protocol version under which each participant is enrolled.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone bromide — Methylnaltrexone will be administered as per the dose and schedule specified in the respective arm.
  Arms: MNTX
Drug: Placebo — Placebo matching to methylnaltrexone will be administered as per the dose and schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and activity of MNTX in relieving opioid-induced constipation following orthopedic procedures.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel-group, placebo- controlled Phase 2 study to evaluate the safety and activity of subcutaneous (SC) MNTX versus SC placebo in participants who have undergone orthopedic procedures and who are expected to require opioids for 1 week after randomization. Participants will sign an informed consent form and be screened between Days 4-10 after their orthopedic procedure. Those participants who meet all eligibility requirements will be enrolled in the study. Treatment with study medication will be continued until either the participant no longer requires opioid medication for pain relief or the maximum number of doses is reached. Originally, participants were receiving treatment for up to 7 days. Then after Protocol Amendment 1 (12 March 2008), the duration of treatment changed from "up to 7 days" to "up to 4 days".

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants greater than or equal to (>=) 18 years of age.
2. Participants must have undergone an orthopedic procedure (that is, total knee or hip replacement, spinal fusion, or reduction of fracture(s) with or without surgical fixation post trauma).
3. Participants must be receiving opioid analgesics (a mu agonist only-not to include agents with mixed mechanisms of action such as tramadol or buprenorphine) after the procedures and be expected to require daily opioid analgesics for at least 7 days post randomization.
4. Participants must be acutely constipated following their orthopedic procedure.
5. Participants must receive all doses of study drug in either hospitals or rehabilitation facilities.
6. Participants must sign an informed consent form.
7. Females of childbearing potential must have a negative pregnancy test and use appropriate birth control throughout the study.
8. Body weight within range of 40 kilograms (kg) - 150 kg (88 - 330 pounds [lbs]).

Exclusion Criteria:

1. Participants with known hypersensitivity to methylnaltrexone, naltrexone, or naloxone.
2. Participants who received any investigational new drug (experimental) in the previous 30 days.
3. Participants who have received a laxative (for example, lactulose) or an enema within 48 hours prior to the first dose.
4. Participants with constipation not attributed to post procedure opioids.
5. Participants with a history of alcohol or prescription or non-prescription drug abuse within the past 2 years.
6. Female participants who are pregnant or lactating.
7. Participants with a known history of chronic active hepatitis B or hepatitis C virus or human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-10-19 (Actual); Primary Completion 2009-01-21 (Actual); Study Completion 2009-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc, Tarrytown, New York, United States

REFERENCES:
- [Derived] Anissian L, Schwartz HW, Vincent K, Vincent HK, Carpenito J, Stambler N, Ramakrishna T. Subcutaneous methylnaltrexone for treatment of acute opioid-induced constipation: phase 2 study in rehabilitation after orthopedic surgery. J Hosp Med. 2012 Feb;7(2):67-72. doi: 10.1002/jhm.943. Epub 2011 Oct 13. PMID 21998076
- See also: Related Info — http://www.progenics.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were randomized in 1:1 ratio to receive either methylnaltrexone (MNTX) or placebo. Originally, participants were receiving treatment for up to 7 days. Then, after Protocol Amendment 1 (12 March 2008), the duration of treatment was changed from "up to 7 days" to "up to 4 days".
Groups:
- MNTX: Participants received methylnaltrexone (MNTX) 12 milligrams (mg) subcutaneously (SC) once daily for up to 4 or 7 days, depending upon the protocol version under which each participant was enrolled.
- Placebo: Participants received placebo matched to MNTX SC once daily for up to 4 or 7 days, depending upon the protocol version under which each participant was enrolled.
Period: Overall Study
Arm/Group | MNTX | Placebo
Started | 19 | 18
Received at Least 1 Dose of Study Drug (Modified intent-to treat (MITT)/Safety population) | 18 | 15
Completed | 15 | 12
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Randomized but not treated | 1 | 3

BASELINE CHARACTERISTICS:
Population: MITT population included all randomized participants who received at least 1 dose of study drug.
Groups:
- MNTX: Participants received MNTX 12 mg SC once daily for up to 4 or 7 days, depending upon the protocol version under which each participant was enrolled.
- Total: Total of all reporting groups
Arm/Group | MNTX | Placebo | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.04) | 65.2 (11.56) | 64.7 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Laxation Response Within 2 Hours of the First Dose
Description: Percentage of participants who had a laxation (that is, bowel movement) within 2 hours after the first dose of study drug, were reported. Participants taking stool softeners within 24 hours of study drug dosing and participants taking rescue laxative medications within 48 hours of study drug dosing were assessed as treatment failures.
Time Frame: 2 hours
Population: MITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MNTX | Placebo
Number analyzed (Participants) | 18 | 15
percentage of participants | 33.33 [13.34 to 59.01] | 0 [0.00 to 0.00]
Statistical Analysis 1: Comparison: MNTX vs Placebo; Analysis was performed using Fisher exact test comparing the percentage of participants with a laxation response within 2 hours of the first dose of study drug, testing MNTX against placebo; Test type: Other; p = 0.0213, Fisher Exact

2. Primary Outcome: Percentage of Participants With Laxation Response Within 4 Hours of the First Dose
Description: Percentage of participants who had a laxation (that is, bowel movement) within 4 hours after the first dose of study drug, were reported. Participants taking stool softeners within 24 hours of study drug dosing and participants taking rescue laxative medications within 48 hours of study drug dosing were assessed as treatment failures.
Time Frame: 4 hours
Population: MITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MNTX | Placebo
Number analyzed (Participants) | 18 | 15
percentage of participants | 38.89 [17.30 to 64.25] | 6.67 [0.17 to 31.95]
Statistical Analysis 1: Comparison: MNTX vs Placebo; Analysis was performed using Fisher exact test comparing the percentage of participants with a laxation response within 4 hours of the first dose of study drug, testing MNTX against placebo; Test type: Other; p = 0.0463, Fisher Exact

3. Secondary Outcome: Time to First Rescue-Free Bowel Movement (Laxation)
Description: A rescue-free laxation was defined as a laxation without use of any rescue medication or rescue procedures. Time to first rescue-free bowel movement following the first dose of study drug was reported.
Time Frame: Baseline (Day 1) up to Day 4 or 7
Population: MITT population included all randomized participants who received at least 1 dose of study drug. One participant with bowel movement prior to dosing was excluded from placebo arm.
Measure: Mean (Standard Error); unit: hours
Arm/Group | MNTX | Placebo
Number analyzed (Participants) | 18 | 14
hours | 23.8 (6.30) | 46.7 (6.49)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Day 30
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | MNTX | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 6/18 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MNTX (N=18) | Placebo (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.